CLINICAL TRIAL: NCT03606408
Title: An Open-label, Multi-center, Roll-over Study to Assess Long Term Safety in Patients With Endogenous Cushing's Syndrome Who Have Completed a Prior Novartis-sponsored Osilodrostat (LCI699) Study and Are Judged by the Investigator to Benefit From Continued Treatment With Osilodrostat
Brief Title: Roll-over Study in Patients With Endogenous Cushing's Syndrome for LCI699
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: RECORDATI GROUP (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLCI699C2X01B
Record Dates: First submitted 2018-07-20; First posted 2018-07-30 (Actual); Results first posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-11

CONDITIONS: Cushing's Syndrome
Keywords: Cushing's syndrome; osilodrostat; LCI699; endogenous Cushing's syndrome
MeSH Terms: conditions — Cushing Syndrome | interventions — Osilodrostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- osilodrostat (Other): open label, with patients receiving same dose as provided in the parent study
  Interventions: Drug: osilodrostat

INTERVENTIONS:
Drug: osilodrostat — osilodrostat, in the form of film coated tablets for oral administration, in the following tablet strengths: 1mg, 5mg, 10mg. Each strength has unique tablet size, colour and imprint.
  Other Names: LCI699

SUMMARY:
The purpose of this study is the evaluation of long-term safety of osilodrostat in patients who have already received osilodrostat treatment in a previous Global Novartis-sponsored trial and who, based on investigators' judgement, will continue benefiting with its administration.

DETAILED DESCRIPTION:
There will be no screening period for this study. Eligible subjects can start their treatment with osilodrostat as soon as they are enrolled in the study. The first study visit will be scheduled at the time of the last study visit for the parent study. Subjects must return to the study center at least on a quarterly basis (every 12 weeks ± 2 weeks) for safety and clinical benefit assessments, and resupply of study medication. Drug dispensing and administration information and adverse events will be collected. The subject may return to the clinic at any given time as per standard of care or treating physician recommendation; however, only the quarterly study visits will be recorded in the Case Report Form (CRF). Study medication dispensed will be recorded in the CRF dose administration page.

All adverse events and serious adverse events, including pregnancy, will be collected throughout the study. Subjects will continue to be treated in this roll-over study until they are no longer benefiting from their osilodrostat treatment as judged by the Investigator or until osilodrostat is commercially available or until one of other discontinuation criteria is met.

ELIGIBILITY:
Inclusion Criteria:

* Patient is currently participating in a Global Novartis-sponsored study receiving osilodrostat for any type of endogenous CS and has fulfilled all their requirements in the parent study.
* Patient is currently benefiting from treatment with osilodrostat, as determined by the Investigator.
* Patient has demonstrated compliance, as assessed by the Investigator, with the parent study protocol requirements.
* Willingness and ability to comply with scheduled visits and treatment plans.
* Written informed consent obtained prior to enrolling into the roll-over study before evaluating the applicability of the subject's participating in the study. -- If consent cannot be expressed in writing, it must be formally documented and witnessed, ideally via an independent trusted witness.

Exclusion Criteria:

* Patient has been permanently discontinued from osilodrostat study treatment in a parent Novartis-sponsor study.
* Patients who are receiving osilodrostat in combination with unapproved or experimental treatments for any type of endogenous CS.
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test. Pregnant or nursing (lactating) women
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing and for 1 week of study after stopping medication. Highly effective contraception methods include:

  * Total abstinence (when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception
  * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy), total hysterectomy, or tubal ligation. at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment
  * Male sterilization (at least 6 months prior to baseline). The vasectomized male partner should be the sole partner for that subject
  * Use of oral, (estrogen and progesterone), injected or implanted hormonal methods of contraception or placement of an intrauterine device (IUD) or intrauterine system (IUS), or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2018-10-05 (Actual); Primary Completion 2023-11-16 (Actual); Study Completion 2023-11-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Recordati, Study Director — Recordati AG
Locations (56):
- United States (10):
  - University of Colorado, Aurora, Colorado
  - Emory University School of Medicine G2304 - C2301, Atlanta, Georgia
  - Northwestern University SC - LCI699C2301, Chicago, Illinois
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Columbia University Medical Center New York Presbyterian Neuroendocrine Unit, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - University of Pennsylvania Medical Center Univ Penn, Philadelphia, Pennsylvania
  - Medical College of Wisconsin MCW 2, Milwaukee, Wisconsin
- Sanatorio Guemes, CABA, Buenos Aires, Argentina
- Universitaetsklinik fuer Innere Medizin III, Vienna, Austria
- Gasthuisberg University Hospital, Leuven, Belgium
- Brazil (4):
  - Universidade Federal do Ceara, Fortaleza, Ceará
  - Hospital Universitario Clementino Fraga Filho, Rio de Janeiro, Rio de Janeiro
  - Hospital do Servidor Publico Estadual de Sao Paulo, São Paulo, São Paulo
  - Hospital das Clinicas da Faculdade de Medicina da USP, São Paulo, São Paulo
- USHATE Akad Ivan Penchev, Sofia, Bulgaria
- Canada (4):
  - University of Alberta Hospital, Edmonton, Alberta
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - Centre de recherche du CHUM CRCHUM, Montreal, Quebec
  - CHUS Hopital Fleurimont, Sherbrooke, Quebec
- China (4):
  - The First Affiliated Hopsital, Sun Yat-Sun University, Guangzhou, Guangdong
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Peking University First Hospital, Beijing
  - Peking Union Medical College Hospital, Beijing
- Clinica Los Yoses, San Pedro, San Jose, Costa Rica, Costa Rica
- France (4):
  - CHU de Bordeaux, Pessac, Cedex
  - Hopital Kremlin Bicetre, Le Kremlin-Bicêtre
  - CHRU de Lille, Lille
  - Hopital Cochin, Paris
- Germany (2):
  - Universitaetsklinikum Erlangen Nuernberg, Erlangen
  - Universitaetsklinikum Muenchen LMU, München
- All India Institute of Medical Sciences, New Delhi, India
- Italy (4):
  - AOU Osp Riuniti Umberto I GM Lancisi G Salesi Univ Studi, Ancona, AN
  - Azienda Ospedaliera di Padova Università degli Studi, Padua, PD
  - Az Ospedaliero Universitaria Pisana Pres Osped di Cisanello, Pisa, PI
  - A O Universitaria Policlinico Federico II Univ Studi Fed II, Napoli
- Japan (2):
  - National Hospital Organization Nagoya Medical Center, Nagoya, Aichi-ken
  - Hyogo College of Medicine Hospital, Nishinomiya, Hyōgo
- Erasmus MC, Rotterdam, Netherlands
- Poland (2):
  - SP ZOZ Szpital Uniwersytecki w Krakowie, Krakow
  - Mazowiecki Szpital Brodnowski, Warsaw
- Center for Endocrinology Russian Academy of Med Sciences, Moscow, Russia
- South Korea (2):
  - Seoul National University Hospital, Seoul
  - Yonsei Univ Health System YUCM, Seoul
- Spain (4):
  - Hospital Universitario Virgen del Rocio, Seville, Andalusia
  - Complejo Uni. Hosp. A Coruña ( antes Hospital Juan Canalejo), A Coruña, Galicia
  - Hospital Gregorio Maranon, Madrid
  - Hospital Universitario i Politecnico La Fe, Valencia
- Thailand (3):
  - King Chulalongkorn Memorial Hospital, Bangkok
  - Siriraj Hospital, Bangkok
  - Songklanagarind Hospital Endocrinology and Metabolism, Songkhla
- Turkey (Türkiye) (3):
  - Istanbul University Cerrahpasa Faculty of Medicine, Istanbul, TUR
  - Marmara University Medical Faculty, Altunizade
  - Kocaeli University Medical Faculty, Kocaeli

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There was no screening period for the study, eligible patients were able to start study treatment as soon as they were enrolled. The study was conducted for 5 years from first patient first visit. Patients continued to be treated in this roll-over study until they no longer received clinical benefit from treatment with osilodrostat (as judged by the Investigator), until osilodrostat was commercially available in their country, or until one of the other discontinuation criteria were met.
Pre-assignment Details: The starting dose of this roll-over study was the same as the one the patients were taking at the end of the parent studies. In addition, they underwent to dose adjustment according to the urine cortisol level and possible AEs. The daily dosage ranged from 1mg every 3 days to 30mg twice a day. So it is not feasible to report the results according to the drug dosage and data has been analysed as one arm.
Groups:
- Osilodrostat: Phase IIb open label, with patients receiving same dose as provided in the parent study
  osilodrostat: osilodrostat, in the form of film coated tablets for oral administration, in the following tablet strengths: 1mg, 5mg, 10mg. Each strength has unique tablet size, colour and imprint.
Period: Overall Study
Arm/Group | Osilodrostat
Started | 127
Completed | 99
Not Completed | 28
Not completed — Adverse Event | 13
Not completed — Withdrawal by Subject | 7
Not completed — Physician Decision | 4
Not completed — Lack of Efficacy | 2
Not completed — Death | 1
Not completed — new therapy for study indication | 1

BASELINE CHARACTERISTICS:
Population: The starting dose of this roll-over study was the same as the one the patients were taking at the end of the parent studies. In addition, they underwent to dose adjustment according to the urine cortisol level and possible AEs. The daily dosage ranged from 1mg every 3 days to 30mg twice a day. So it is not feasible to report the results according to the drug dosage and data has been analysed as one arm.
Arm/Group | Osilodrostat
Number analyzed (Participants) | 127
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.2 (12.39)
Age, Customized [Count of Participants; unit: Participants]
  <65 years | 119
  ≥65 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 95
  Male | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14
  Not Hispanic or Latino | 94
  Unknown or Not Reported | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 26
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 96
  More than one race | 0
  Unknown or Not Reported | 1
Weight [Mean (Standard Deviation); unit: kg] | 74.59 (21.253)
Height [Mean (Standard Deviation); unit: cm] | 163.73 (9.839)
Body Mass Index [Mean (Standard Deviation); unit: Kg/m^2] | 27.84 (7.631)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse/Serious Adverse Events
Description: To evaluate long-term safety data with osilodrostat treatment (Frequency and severity of adverse events (AEs)/serious adverse events (SAEs))
Time Frame: up to 5 years
Population: The starting dose of this roll-over study was the same as the one the patients were taking at the end of the parent studies. In addition, they underwent to dose adjustment according to the urine cortisol level and possible AEs. The daily dosage ranged from 1mg every 3 days to 30mg twice a day. So, the results are not reported according to the drug dosage and data has been analysed as one arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Osilodrostat
Number analyzed (Participants) | 127
Participants
  Adverse events (AEs) | 115
  Treatment-related AEs | 50
  Adverse events of CTCAE Grade ≥ 3 | 34
  Treatment-related AEs of CTCAE Grade ≥ 3 | 3
  Serious adverse events | 35
  Treatment-related SAEs | 4
  Fatal SAEs | 2
  Treatment-related fatal SAEs | 0
  Adverse events leading to discontinuation | 14
  Treatment-related AEs leading to discontinuation | 5
  Adverse events leading to dose interruption or adjustment | 56
  Treatment-related AEs leading to dose interruption or adjustment | 35
  Adverse events requiring additional therapy | 94
  Treatment-related AEs requiring additional therapy | 17
  Adverse events of special interest (AESIs) | 51
  Treatment-related AESIs | 29

2. Secondary Outcome: Percentage of Patients With Clinical Benefit
Description: Proportion of patients with clinical benefit as assessed by the Investigator at scheduled visits based on medical check-up and lab values such as Urine Free Cortisol.
Time Frame: up to of 5 years
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Osilodrostat
Number analyzed (Participants) | 127
Participants
  Week 1 | 127
  Week 12 | 122
  Week 24 | 119
  Week 36 | 114
  Week 48 | 103
  Week 96 | 74
  Week 144 | 52
  End of treatment | 99

ADVERSE EVENTS:
Time Frame: From enrolment up to 30 days after the last administration of study treatment (up to 5 years)
Description: The starting dose of this roll-over study was the one the patients were taking at the end of the parent studies. In addition, they underwent to dose adjustment according to the UCF and possible AEs. The daily dosage ranged from 1mg every 3 days to 30mg twice a day. The data has been analysed as one arm. Two patients experienced fatal SAEs before the Safety Follow-up, reported under the PTs of COVID-19 and respiratory failure, not related to the disease or treatment
Arm/Group | Osilodrostat
All-Cause Mortality (participants affected / at risk) | 2/127
Serious Adverse Events (participants affected / at risk) | 35/127
Other Adverse Events (participants affected / at risk) | 115/127
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Osilodrostat (N=127)
COVID-19 (Infections and infestations) | 7
Cholelithiasis (Hepatobiliary disorders) | 3
Pitituary tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Adrenal insufficiency (Endocrine disorders) | 2
ACTH-producing pituitary tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Acute stress disorder (Psychiatric disorders) | 1
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Alanine aminotransferase increased (Investigations) | 1
Appendicitis (Infections and infestations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Bile duct stone (Hepatobiliary disorders) | 1
Biliary dilatation (Hepatobiliary disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Device dislocation (Product Issues) | 1
Disease progression (General disorders) | 1
Diverticulitis (Gastrointestinal disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Food poisoning (Gastrointestinal disorders) | 1
Gamma-glutamyl transferase increased (Investigations) | 1
Hand fracture (Injury, poisoning and procedural complications) | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1
Influenza like illness (General disorders) | 1
Liver function test abnormal (Investigations) | 1
Nausea (Gastrointestinal disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Paralysis (Nervous system disorders) | 1
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pituitary-dependent Cushing's syndrome (Endocrine disorders) | 1
Pneumonia (Infections and infestations) | 1
Pneumonia bacterial (Infections and infestations) | 1
Radius fracture (Injury, poisoning and procedural complications) | 1
Renal colic (Renal and urinary disorders) | 1
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Retinal vein thrombosis (Eye disorders) | 1
Ureterolithiasis (Renal and urinary disorders) | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Osilodrostat (N=127)
Hypertension (Vascular disorders) | 11
COVID-19 (Infections and infestations) | 29
Abdominal pain (Gastrointestinal disorders) | 9
Adrenal insufficiency (Endocrine disorders) | 16
Vomiting (Gastrointestinal disorders) | 9
Nausea (Gastrointestinal disorders) | 14
Diarrhoea (Gastrointestinal disorders) | 13
Asthenia (General disorders) | 9
Fatigue (General disorders) | 9
Pyrexia (General disorders) | 8
Nasopharyngitis (Infections and infestations) | 12
Influenza (Infections and infestations) | 11
Upper respiratory tract infection (Infections and infestations) | 10
Urinary tract infection (Infections and infestations) | 7
Cortisol free urine increased (Investigations) | 13
SARs-Cov-2 test positive (Investigations) | 13
Blood corticotrophin increased (General disorders) | 8
Decreased appetite (Metabolism and nutrition disorders) | 9
Back pain (Musculoskeletal and connective tissue disorders) | 11
Arthralgia (Musculoskeletal and connective tissue disorders) | 9
Headache (Nervous system disorders) | 16
Dizziness (Nervous system disorders) | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 7
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (3):
  • Study Protocol (2020-05-06): https://cdn.clinicaltrials.gov/large-docs/08/NCT03606408/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-05): https://cdn.clinicaltrials.gov/large-docs/08/NCT03606408/SAP_001.pdf
  • Informed Consent Form (2022-03-07): https://cdn.clinicaltrials.gov/large-docs/08/NCT03606408/ICF_002.pdf